CLINICAL TRIAL: NCT04974437
Title: Quantitative Assessment of the Activation of Brain Areas With Positive and Negative Emotional Stimuli and Its Correlation With Degrees of Emotional Disorder.
Brief Title: Metabolic Activation of Brain Areas With Emotional Stimuli Compared With Score in Psychological Test
Acronym: fMRI
Status: Completed | Type: Observational
Sponsor: Instituto del Corazon, Argentina (Other)
Responsible Party: Principal Investigator, Ruben Novoa, MD, Head of Magnetic Resonance Imaging, Principal Investigator, Instituto del Corazon, Argentina
Other Study IDs: 2
Record Dates: First submitted 2021-06-23; First posted 2021-07-23 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Emotional Disorder
Keywords: fMRI; Emotion; Cerebral blood volume

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Quantitative assessment of the activation of brain areas by functional magnetic resonance imaging (fRMI) in the face of positive and negative emotional stimuli using audiovisual materials validated for the local population and its correlation with degrees of emotional disorder based on a score obtained by a validated questionnaire for the local population, in 16 volunteers from the city of La Rioja in Argentina.

DETAILED DESCRIPTION:
The technology applied in fMRI allows us to visualize on a color scale the changes in blood flow in those sectors of the brain that increase their metabolic activity during a given action. This is achieved by mapping the cerebral blood volume, which increases or decreases according to the metabolic activity in a certain region of the brain. This indirect method of measuring the metabolic activity of brain areas is very useful for anatomically identifying motor areas and critical functions in individual patients prior to neurosurgery, to allow better surgical planning. Currently this is its main application in healthcare practice. In the field of research it is applied in clinical neurology, psychiatry and psychology. Studies have been conducted on the activations of brain regions in basic emotions. There is less data on the quantitative differences of these activations in the Argentine population according to the degree of emotional disorder, this being the object of study of this project. Emotional disorders are transversal to different pathologies, with or without a psychotic component.

ELIGIBILITY:
Inclusion Criteria:

- Must be able to understand the instructions and collaborate during the data adquisition.

Exclusion Criteria:

* Any contraindication to enter an MRI (for example, a pacemaker)
* Claustrophobia.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer participants from the population of the city of La Rioja in Argentina, over 21 years of age.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Differences in fMRI brain activation response in specific brain regions in response to positive and negative emotional stimuli | Cross sectional adquistion of data with fMRI in a 20 minutes session after answering a questionnaire.
  A score will be assigned to each participant according to the results obtained in a validated questionnaire to categorize emotional disorder with 37 questions, each of them with a score of 0, 1 or 2 according to the answer, to give a score to each participant that will be on the scale from 0 to 74.
  The stimuli consist of the projection of audiovisual material validated to generate positive or negative emotions. The activations are quantified in a 1.5 Tesla resonator and the units of measurement for each region of interest will be cm3 of activated tissue and Z-value of fMRI activation.
  Once the informed consent is signed, the participant is asked to answer the questionnaire to categorize the emotional score. After this survey, the fMRI is acquired, measuring the activation by areas from the beginning of the audiovisual stimuli until their completion. The time for the fMRI acquisition session for each participant in this cross-sectional study is estimated 20-minute .

CONTACTS AND LOCATIONS:
Overall Officials: Ruben F Novoa, MD, Principal Investigator — InCor Heart Institute
Locations (1):
- Incor, La Rioja, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices) will be shared with researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication and ending 36 months following article publication.
Access Criteria: Proposals should be directed to rubennnovoa@gmail.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Michelini, Y. Características de la experiencia emocional inducida mediante fragmentos de películas en una muestra de jóvenes argentinos. Interdisciplinaria, 2015, 32, 2, 367-382.
- [Background] Muñoz Rodriguez M, Korzeniowski C. Validación del cuestionario epidemiológico en sintomatología mental -CESIM- en población Argentina. Revista de Salud Pública, (XXIII) 2:8-24 Junio 2019
- [Background] Gu S, Wang F, Cao C, Wu E, Tang YY, Huang JH. An Integrative Way for Studying Neural Basis of Basic Emotions With fMRI. Front Neurosci. 2019 Jun 19;13:628. doi: 10.3389/fnins.2019.00628. eCollection 2019. PMID 31275107
- [Background] Kragel PA, Knodt AR, Hariri AR, LaBar KS. Decoding Spontaneous Emotional States in the Human Brain. PLoS Biol. 2016 Sep 14;14(9):e2000106. doi: 10.1371/journal.pbio.2000106. eCollection 2016 Sep. PMID 27627738
- [Background] Kragel PA, LaBar KS. Multivariate neural biomarkers of emotional states are categorically distinct. Soc Cogn Affect Neurosci. 2015 Nov;10(11):1437-48. doi: 10.1093/scan/nsv032. Epub 2015 Mar 25. PMID 25813790
- [Background] Kassam KS, Markey AR, Cherkassky VL, Loewenstein G, Just MA. Identifying Emotions on the Basis of Neural Activation. PLoS One. 2013 Jun 19;8(6):e66032. doi: 10.1371/journal.pone.0066032. Print 2013. PMID 23840392
- [Background] Gur RE, Gur RC. Functional magnetic resonance imaging in schizophrenia. Dialogues Clin Neurosci. 2010;12(3):333-43. doi: 10.31887/DCNS.2010.12.3/rgur. PMID 20954429
- [Background] Posner J, Russell JA, Gerber A, Gorman D, Colibazzi T, Yu S, Wang Z, Kangarlu A, Zhu H, Peterson BS. The neurophysiological bases of emotion: An fMRI study of the affective circumplex using emotion-denoting words. Hum Brain Mapp. 2009 Mar;30(3):883-95. doi: 10.1002/hbm.20553. PMID 18344175
- [Background] Rios-Lago M. [Functional magnetic resonance and neuropsychology: basic concepts]. Radiologia. 2008 Sep-Oct;50(5):351-65; quizz 365. doi: 10.1016/s0033-8338(08)76050-8. Spanish. PMID 19055911

DOCUMENTS (2):
  • Study Protocol (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT04974437/Prot_002.pdf
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT04974437/ICF_001.pdf